CLINICAL TRIAL: NCT04132765
Title: Reliability and Construct Validity of the Turkish Version of the Drooling Impact Scale Among Children With Cerebral Palsy
Brief Title: Turkish Validation of The Drooling Impact Scale
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2019.963
Record Dates: First submitted 2019-10-17; First posted 2019-10-21 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-10

CONDITIONS: Hypersalivation; Cerebral Palsy
Keywords: cerebral palsy; drooling impact scale; hypersalivation; validity
MeSH Terms: conditions — Sialorrhea; Cerebral Palsy | interventions — Eating

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with cerebral palsy: Patients with cerebral palsy at between the ages of 4-16 years and at Gross Motor Function Classification Levels of 3,4,5
  Interventions: Other: Drooling Impact Scale; Other: Drooling Frequency and Severity Scale; Other: The Caregiver Priorities and Child Health Index of Life with Disabilities (CPCHILD™); Other: Drooling Quotient (DQ); Other: Patient and caregiver visual analog scale (VAS) for drooling; Other: Functional Oral Intake Scale (FOIS); Other: number of bibs daily used; Other: number of hospital admissions per year related to respiratory infections; Other: Gross Motor Function Classification System (GMFCS); Other: Manual Ability Classification System (MACS); Other: Communication Function Classification System (CFCS); Other: Eating and Drinking Ability Classification System (EDACS)

INTERVENTIONS:
Other: Drooling Impact Scale — A scale with 10 items which are scored with visual analog scale from1 to 10. Drooling impact increases with increased scores.
Other: Drooling Frequency and Severity Scale — In this scale, parents or care givers were asked to rate the severity and frequency of drooling, classifying severity of drooling using a 5-level domain ranging from 1 (dry) to 5 (profuse drooling). The frequency of drooling was classified using a 4-level domain ranging from 1(no drooling) to 4 (constant drooling)
Other: The Caregiver Priorities and Child Health Index of Life with Disabilities (CPCHILD™) — A quality of life scale that measure caregivers' perspectives on the health status, comfort, well being, and ease of caregiving of children with severe developmental disabilities. CPCHILD consists of 36 items distributed over six sections representing the following domains: (1) Personal Care (eight items); (2) Positioning, Transfer, and Mobility (eight items); (3) Communication and Social Interaction (seven items); (4) Comfort, Emotions, and Behaviour (nine items); (5) Health (three items); and (6) Overall Quality Of Life (one item). For the sections which involve the performance of skills, the degree of difficulty of accomplishing each task or activity was rated on a 7-point ordinal scale anchored by 0 ('No problem at all') to 6 ('Impossible').
Other: Drooling Quotient (DQ) — DQ is a semi-quantitative method that assesses the presence of newly formed saliva on the lips every 15 seconds with 40 observations in 10 minutes, expressed as a percentage based on the ratio between the number of observed drooling episodes and the total number of observations.
Other: Patient and caregiver visual analog scale (VAS) for drooling — Patients will be asked to score their children's drooling severity on a visual analog scale (0-100 mm, 0 none to 100 severe)
Other: Functional Oral Intake Scale (FOIS) — Functional Oral Intake Scale (FOIS) which is a 7-point ordinal scale document the functional level of oral intake of food and liquid.
Other: number of bibs daily used — Parents will be asked their children's number of bibs daily used.
Other: number of hospital admissions per year related to respiratory infections — Parents will be asked their children's number of hospital admissions per year related to respiratory infections.
Other: Gross Motor Function Classification System (GMFCS) — The GMFCS describes self-initiated movement and use of assistive devices (walkers, crutches, canes, wheelchairs) for mobility during an individual's usual activity.
Other: Manual Ability Classification System (MACS) — The MACS is also a simple, five-point ordinal classification system and was designed for use in children ages 4-18 years. The MACS is a validated measure in cerebral palsy that can be used to classify a child's typical use of both hands and upper limbs.
Other: Communication Function Classification System (CFCS) — The CFCS is a simple, five-point ordinal classification system that assesses everyday communication (not optimal communication) of children with cerebral palsy.
Other: Eating and Drinking Ability Classification System (EDACS) — EDACS is a measure to assess eating and drinking ability for children with CP, ages 3 and older. This classification is a simple five-point ordinal system.

SUMMARY:
The aim of this study is to investigate the reliability and construct validity of the Turkish version of the Drooling Impact Scale in children with cerebral palsy

DETAILED DESCRIPTION:
Drooling is common among several neurologic disorders such as cerebral palsy, Parkinson's disease, amyotrophic lateral sclerosis, which are the main diseases that physiatrist are one of the leading physicians involved in whose management 1. Drooling can be seen either as anterior drooling, unintentional leaving of saliva from mouth to outside of the body, or posterior drooling, invisible spill of saliva from mouth through pharyngeal isthmus and then to respiratory or digestive tract, inside the body 2. Anterior drooling causes psycho-social impairment, skin problems, infections, bad odor, dehydration, dentation problems and wet clothes and tools while posterior drooling may result in morbidity by posing a risk for aspiration pneumonia. Despite the frequency and significance of the condition, there is still a paucity of research and inadequate evidence about the various treatments and valid and reliable outcomes available. A major problem for research into interventions to reduce drooling is that there is no valid and reliable measurement tool of saliva control. There is no questionnaire in Turkish to evaluate the effects of drooling as well as drooling interventions.The aim of this study is to investigate the reliability and construct validity of the Turkish version of the Drooling Impact Scale in children with cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unilateral or bilateral cerebral palsy at between the ages of 4-16
2. Spastic, dyskinetic or mixed type cerebral palsy
3. GMFCS level 3,4,5
4. Stable drooling within at least one month

Exclusion Criteria:

1. Active infection of salivary glands
2. Upper respiratory tract infection at the time of testing
3. History of anticholinergic drug intake in the past three weeks
4. Occurance of any above between test and re-test assessment that may interfere with the results

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with unilateral or bilateral, spastic, dyskinetic or mixed type cerebral palsy at between the ages of 4-16 and GMFCS level 3,4,5
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-11-25 (Actual); Primary Completion 2020-08-30 (Estimated); Study Completion 2020-08-30 (Estimated)

PRIMARY OUTCOMES:
Drooling Impact Scale | Day 0
  A scale with 10 items which are scored with visual analog scale from1 to 10. Drooling impact increases with increased scores.
Drooling Impact Scale | Day 3
  A scale with 10 items which are scored with visual analog scale from1 to 10. Drooling impact increases with increased scores.

SECONDARY OUTCOMES:
Drooling Frequency and Severity Scale | Day 0
  n this scale, parents or care givers were asked to rate the severity and frequency of drooling, classifying severity of drooling using a 5-level domain ranging from 1 (dry) to 5 (profuse drooling). The frequency of drooling was classified using a 4-level domain ranging from 1(no drooling) to 4 (constant drooling)
The Caregiver Priorities and Child Health Index of Life with Disabilities (CPCHILD™) | Day 0
  A quality of life scale that measure caregivers' perspectives on the health status, comfort, well being, and ease of caregiving of children with severe developmental disabilities. CPCHILD consists of 36 items distributed over six sections representing the following domains: (1) Personal Care (eight items); (2) Positioning, Transfer, and Mobility (eight items); (3) Communication and Social Interaction (seven items); (4) Comfort, Emotions, and Behaviour (nine items); (5) Health (three items); and (6) Overall Quality Of Life (one item). For the sections which involve the performance of skills, the degree of difficulty of accomplishing each task or activity was rated on a 7-point ordinal scale anchored by 0 ('No problem at all') to 6 ('Impossible').
Drooling Quotient (DQ) | Day 0
  DQ is a semi-quantitative method that assesses the presence of newly formed saliva on the lips every 15 seconds with 40 observations in 10 minutes, expressed as a percentage based on the ratio between the number of observed drooling episodes and the total number of observations.
Patient and caregiver visual analog scale (VAS) for drooling | Day 0
  Patients will be asked to score their children's drooling severity on a visual analog scale.
Functional Oral Intake Scale (FOIS) | Day 0
  Functional Oral Intake Scale (FOIS) which is a 7-point ordinal scale document the functional level of oral intake of food and liquid.
number of bibs daily used | Day 0
  Parents will be asked their children's number of bibs daily used.
number of hospital admissions per year related to respiratory infections | Day 0
  Parents will be asked their children's number of hospital admissions per year related to respiratory infections.
Gross Motor Function Classification System (GMFCS) | Day 0
  The GMFCS describes self-initiated movement and use of assistive devices (walkers, crutches, canes, wheelchairs) for mobility during an individual's usual activity.
Manual Ability Classification System (MACS) | Day 0
  The MACS is also a simple, five-point ordinal classification system and was designed for use in children ages 4-18 years. The MACS is a validated measure in cerebral palsy that can be used to classify a child's typical use of both hands and upper limbs.
Communication Function Classification System (CFCS) | Day 0
  The CFCS is a simple, five-point ordinal classification system that assesses everyday communication (not optimal communication) of children with cerebral palsy.
Eating and Drinking Ability Classification System (EDACS) | Day 0
  EDACS is a measure to assess eating and drinking ability for children with CP, ages 3 and older. This classification is a simple five-point ordinal system.

CONTACTS AND LOCATIONS:
Overall Officials: Evrim Karadag Saygi, Prof, Study Chair — Marmara University; Nida Yektauşakları, PT, Principal Investigator — Marmara University School of Health Sciences; Fatma Özer, Student, Principal Investigator — Marmara University
Locations (1):
- Esra Giray, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study will be available on request from the corresponding author (EG). The data will not be publicly available due to their containing information that could compromise the privacy of research participants.

REFERENCES:
- [Result] Lakraj AA, Moghimi N, Jabbari B. Sialorrhea: anatomy, pathophysiology and treatment with emphasis on the role of botulinum toxins. Toxins (Basel). 2013 May 21;5(5):1010-31. doi: 10.3390/toxins5051010. PMID 23698357
- [Result] Erasmus CE, van Hulst K, Rotteveel JJ, Willemsen MA, Jongerius PH. Clinical practice: swallowing problems in cerebral palsy. Eur J Pediatr. 2012 Mar;171(3):409-14. doi: 10.1007/s00431-011-1570-y. Epub 2011 Sep 20. PMID 21932013
- [Result] Pesheva P, Kuklinski S, Schmitz B, Probstmeier R. Galectin-3 promotes neural cell adhesion and neurite growth. J Neurosci Res. 1998 Dec 1;54(5):639-54. doi: 10.1002/(SICI)1097-4547(19981201)54:53.0.CO;2-2. PMID 9843155
- See also: Sialorrhea: A Guide to Etiology, Assessment, and Management — https://www.researchgate.net/publication/330749140_Sialorrhea_A_Guide_to_Etiology_Assessment_and_Management